CLINICAL TRIAL: NCT06399627
Title: Effect of Non-anemic Iron Deficiency on Outcome Following Off-pump Coronary Revascularization
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-1112
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Bypass, Off-Pump; Iron Deficiencies
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Iron replete: Patient who did not meet the criteria for iron deficiency (see below)
- Iron deficient: patients with preoperative iron profile of either of the following were defined as iron deficient:
  1. serum ferritin <100mcg/L
  2. 100mcg/L < serum ferritin <300mcg/L and
     * transferrin saturation < 20% or
     * C reactive protein ≥ 5mg/L

SUMMARY:
This is a single center retrospective study of patients who underwent off pump coronary artery bypass surgery between 2016.11~2023.05. From this patient group, preoperatively non-anemic patients were selected and were divided into 2 cohorts according to their preoperative iron status; iron replete and iron deficient. These two cohorts were compared to evaluate the effect of preoperative iron deficiency on patient outcomes.

The primary end point was the occurrence of composite morbidity/mortality end points which were: in hospital mortality, acute kidney injury (AKI), stroke, deep sternal infection, hemostatic reoperation, prolonged mechanical ventilation of more than 24hours, delirium and postoperative myocardial infarction. Occurrence of any one of these outcomes counted as primary end point met. Secondary outcome was to evaluate and compare hemoglobin recovery of iron replete and deficient patients until one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received off pump coronary artery bypass surgery (OPCAB) between 2016.11.01-2023.05.31

Exclusion Criteria:

* preoperative anemia (male Hb <13g/dL, female Hb<12g/dL)
* emergency surgery
* redo-off pump coronary artery bypass surgery
* minimally invasive coronary artery bypass surgery
* OPCAB in conjunction with other cardiac surgical procedures (e.g. valve surgery, graft replacement surgery of the aorta)
* intraoperative on pump conversion
* lack of sufficient preoperative data (ferritin, transferrin saturation, C-reactive protein) to determine iron status
* administration of intravenous iron within 4 weeks or parenteral iron of more than 2 weeks prior to surgery
* enrollemnt in other clinical studies

Ages: 29 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-anemic patients who underwent off pump coronary artery bypass surgery
Sampling Method: Probability Sample
Enrollment: 433 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with in hospital mortality, stroke, deep sternal infection, hemostatic reoperation, delirium | from the end of surgery until patient discharge (assessed up to day 60)
  This outcome is a composite of the following: in hospital mortality, acute kidney injury (AKI), stroke, deep sternal infection, hemostatic reoperation, prolonged mechanical ventilation of more than 24hours, delirium and postoperative myocardial infarction. The occurrence of any one of these was regarded as primary end point met.
Number of participants with acute kidney injury | until 7 days after surgery
  This outcome is a composite of the following: in hospital mortality, acute kidney injury (AKI), stroke, deep sternal infection, hemostatic reoperation, prolonged mechanical ventilation of more than 24hours, delirium and postoperative myocardial infarction. The occurrence of any one of these was regarded as primary end point met.
Number of participants with post operative myocardial infarction | until 48 hours post-surgery
  This outcome is a composite of the following: in hospital mortality, acute kidney injury (AKI), stroke, deep sternal infection, hemostatic reoperation, prolonged mechanical ventilation of more than 24hours, delirium and postoperative myocardial infarction. The occurrence of any one of these was regarded as primary end point met.

SECONDARY OUTCOMES:
Post discharge hemoglobin | Until 1 year after surgery
  Data of hemoglobin levels after discharge until 1 year after surgery was collected to evaluate hemoglobin recovery to preoperative baseline levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health system, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No